CLINICAL TRIAL: NCT01742858
Title: Establishment of Normative Data of Brain Network Activation Analysis (BNA) Using Evoked Response Potentials, in Adolescents and Young Adults
Brief Title: Normative Data of Brain Network Activation
Status: Withdrawn | Type: Observational
Why Stopped: The study was halted due to logistical reasons.
Sponsor: ElMindA Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: ELM-07
Record Dates: First submitted 2012-12-03; First posted 2012-12-06 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Healthy Controls

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Adolescents: 15-18 years old
- Young adults I: 19-24 years old
- Young adults II: 25-30 years old

SUMMARY:
Establish normative data of ElMindA's Brain Network Activation (BNA) using evoked response in three age groups.

DETAILED DESCRIPTION:
Currently, there is no reliable, bedside, and non-invasive method for assessing connectivity changes in electrophysiological activity of the brain associated with brain-related pathologies, e.g., concussion, ADHD, autistic spectrum disorders (ASD), etc. Event Related Potentials (ERPs), which are temporal reflections of the neural mass electrical activity of cells in specific regions of the brain that occur in response to stimuli, may offer such a method, as they provide both a non-invasive and portable measure of brain function. The ERPs provide excellent temporal information, but spatial resolution for ERPs has traditionally been limited. However, by using high-density electroencephalograph (EEG) recording spatial resolution for ERPs is improved significantly. The paradigm for the current study will combine neurophysiological knowledge with mathematical signal processing and pattern recognition methods (BNA) to temporally and spatially map brain function, connectivity and synchronization.

The need of objective measures that will help the clinician in its decision making in brain-related pathologies is recognized. BNA is a new imaging modality that has been developed to fill this gap.

ELIGIBILITY:
Inclusion Criteria:

* Age 15-30 years.
* Able to speak, read and understand English sufficiently to understand the nature of the study, and to allow completion of all study assessments.
* Willingness to participate and able to give informed assent (child) and/or consent (parent for minors or adult 18+ years of age for self).

Exclusion Criteria:

* Currently participate in a contact sport (e.g., football, hockey, soccer, rugby, lacrosse, martial arts).
* Currently with lice or open wounds on scalp.
* Any chronic disease as determined by clinical evaluation and medical history.
* Any psychiatric disorder, e.g., depression, bipolar disorder, schizophrenic disorder, etc. as determined by clinical evaluation and the Mini International Neuropsychiatric Interview (MINI)
* Any CNS neurologic disorder, e.g., epilepsy, seizures, etc. as determined by clinical evaluation
* History of Special education, e.g., reading disorder (dyslexia), writing disorder (dysgraphia), math disorder (dyscalculia), nonverbal learning disorder.
* History of any medication affecting CNS within the last 3 months, e.g., antidepressants, anticonvulsants, psychostimulants, first generation antihistamines, etc.
* Substance abuse in the last 3 months.
* Significant sensory deficits, e.g., deafness or blindness.
* History of any clinically significant brain trauma as determined by the investigator

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Experimental subjects will include males and females recruited from the Eugene metropolitan area.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-02; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Functional networks of brain activity in healthy individuals measured using analysis of EEG Event Related Potential (ERP) data | 1 week
  The study outcome measure are functional networks of brain activity of healthy adolescents (age 15-18 years) and young adults (19-24, 25-30 years) established based on an analysis of EEG data recorded while study subjects perform ERP tasks

CONTACTS AND LOCATIONS:
Overall Officials: Don Tucker, PhD, Principal Investigator — Electrical Geodesics, Inc.
Locations (1):
- Electrical Geodesics, Inc., Eugene, Oregon, United States